CLINICAL TRIAL: NCT06581133
Title: Introducing a Structured Sleep Disruption Pattern to Provoke Earlier Seizures During Epilepsy Monitoring Unit Admissions
Brief Title: Sleep Disruption Pattern - Epilepsy Monitoring Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00115255
Record Dates: First submitted 2024-04-04; First posted 2024-09-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy Intractable
Keywords: epilepsy monitoring unit
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: During their epilepsy monitoring unit (EMU) admission, patients will be divided into either the alarm group or the control group. Patients in the alarm group will have an alarm system placed in their room, scheduled to sound at several timepoints during the night. This intervention will be conducted throughout the whole EMU admission. Patients in the control group will have an alarm system placed in their room, but the alarm system will not sound during any of the nights during their EMU admission.
Who Masked: Participant
Masking Description: This is a single blind study and patients will not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alarm (Experimental): Patients in the alarm group will have an alarm system placed in their room, scheduled to sound at 4 timepoints during the night (specific timepoints adjusted based on patient's preferred bed times). This intervention will stop when the clinical team has collected sufficient seizures for clinical decision making.
  Interventions: Device: Alarm system
- Control (No Intervention): Patients in the control group will have an alarm system placed in their room, but the alarm system will not sound during any of the nights during their EMU admission.

INTERVENTIONS:
Device: Alarm system — Generic alarm system programmed to sound during the night to try to induce arousals from sleep.
  Arms: Alarm

SUMMARY:
Epilepsy affects millions worldwide, with 40% of patients experiencing uncontrolled seizures despite medication. Comprehensive epilepsy centers recommend continuous video-electroencephalography monitoring to define seizure type and distinguish mimickers. This process, however, is resource-intensive, with lengthy hospital stays. The investigators' recent study identified a heightened association between arousals and epileptic activity in drug-resistant focal epilepsy patients. Building on these findings, the investigators aim to explore whether disrupting sleep with an alarm system triggers earlier occurrence of seizures, potentially offering insights to reduce hospital stay durations in epilepsy monitoring units.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to 60 years
* EMU monitoring for presurgical evaluations
* Average 2-3 seizures per week based on pre-admission seizure diary
* Sleep as a known seizure trigger

Exclusion Criteria:

- Multiple seizures a day based on pre-admission seizure diary

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency during EMU (epilepsy monitoring unit) stay | 1 month after the EMU stay (up to 9 weeks)
  Average number of seizures per day, recorded daily during the patient's EMU stay. Measured for all groups of patients.
Duration of EMU (epilepsy monitoring unit) admission | 1 month after the EMU stay (up to 9 weeks)
  Overall duration (in days) of the EMU admission. Measured for all groups of patients.
Average interictal spike rates | 1 month after the EMU stay (up to 9 weeks)
  Average number of spike rates, taken from a random segment for each day and night. Measured for all groups of patients.
Change in sleep quality | Baseline (Day 1), last day of EMU stay (up to 5 weeks), 1 month after the EMU stay (up to 9 weeks)
  As determined by changes in Pittsburgh Sleep Quality Index scores. A higher score indicates increased sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Frauscher, MD PD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No